CLINICAL TRIAL: NCT01177020
Title: The Role of Pro-angiogenic Immune Cells in Human Pregnancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Elad Mei-Dan, MD, Hillel Yaffe Medical Center
Other Study IDs: HYMC1069A
Record Dates: First submitted 2010-05-12; First posted 2010-08-06 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-08

CONDITIONS: Fetal Growth Retardation; Preeclampsia
MeSH Terms: conditions — Fetal Growth Retardation; Pre-Eclampsia | interventions — Biological Specimen Banks

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Placentas after delivery or abortion
  Interventions: Other: Biological specimen

INTERVENTIONS:
Other: Biological specimen — Biological specimen taken from placenta

SUMMARY:
Identification of the presence of proangiogenic immune cells in normal human placentas may enable predication of some pregnancy disorders.

ELIGIBILITY:
Inclusion Criteria:

* Placentas that have been delivered in the Medical Center

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Placentas after delivery or abortion
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To find the angiogenic potential of proangiogenic immune cells derived from human placentas. | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel